CLINICAL TRIAL: NCT05875363
Title: Neurodevelopmental Disorders in Youth With Criminal Behaviors
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202103130RIND
Record Dates: First submitted 2023-04-13; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Autistic Spectrum Disorder; Conduct Disorders in Adolescence
Keywords: neurodevelopmental disorder; criminality; adolescence
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Neurodevelopmental Disorders; Criminal Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ADHD: ADHD is among the most commonly diagnosed neurodevelopmental disorders, and the worldwide prevalence.
  Interventions: Other: collect data
- ASD: Autistic spectrum disorder (ASD), characterized by overriding obsessions and difficulties in social cognition, might render the affected individuals vulnerable for becoming an offender or a victim of crime.
  Interventions: Other: collect data
- Other disorders in youth: CD or substance use disorder: Conduct disorder (CD), characterized by antisocial and aggressive behavior, affects 2-2.5% of children and adolescents. CD is a risk factor for antisocial personality disorder, and despite the fact that a CD diagnosis completely relies on behavioral symptoms, research has identified neurocognitive impairments.
  Interventions: Other: collect data

INTERVENTIONS:
Other: collect data — The Juvenile Affairs Division provided the records without person-identifiable data (i.e., name, ID) to the researchers. The researchers coded the above data (i.e., the offenders' sociodemographic data, medical history, and criminal history).
  Demographic characteristics were collected, which are the offenders' age, gender, occupation, education level, and residence (district). We recorded the offenders' household members (without the name or age), main caregivers (e.g., father, or mother), and the parents' socioeconomic and marital status. We also tracked whether the offenders live with family members with mental illness, whether they are from at-risk families, and whether had been victims of domestic violence. The medical history and deviant (or criminal) behaviors will be collected in the attached measure.

SUMMARY:
1. Describe the prevalence of neurodevelopmental disorders among youth with criminal behaviors
2. Explore the relationship between specific neurodevelopmental disorders and the rates and types of crime
3. Examine the roles of psychiatric comorbidities and sociodemographic factors in juvenile criminality

ELIGIBILITY:
Inclusion Criteria:

* Juvenile offender from The Juvenile Affairs Division of Taipei City Police Department

Exclusion Criteria:

* Not Juvenile offender

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This retrospective study is based on the counseling registry of the Juvenile Affairs Division of Taipei City Police Department. The dataset encompasses around 1000 juvenile offenders who were actively followed up by the counselors of the division. The records include the offenders' sociodemographic data, medical history, and criminal history without person-identifiable data (i.e., name, ID).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of ADHD, ASD, and other neurodevelopmental disorder in juvenile offender | 3 years
  Statistical analysis done by SAS (v.9.4) examine the prevalence of each neurodelopmental disorder, such as ADHD and ASD.
Age of first criminal behavior | 3 years
  Based on different neurodevelopmental disorder diagnosis, determine whether the data is able to predict onset and type of criminal behaviors for each juvenile offender.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The collected data only stay in Dr.Chien's lab

REFERENCES:
- [Background] Moore KE, Oberleitner LMS, Zonana HV, Buchanan AW, Pittman BP, Verplaetse TL, Angarita GA, Roberts W, McKee SA. Psychiatric Disorders and Crime in the US Population: Results From the National Epidemiologic Survey on Alcohol and Related Conditions Wave III. J Clin Psychiatry. 2019 Feb 12;80(2):18m12317. doi: 10.4088/JCP.18m12317. PMID 30758921
- [Background] Lamberti JS, Katsetos V, Jacobowitz DB, Weisman RL. Psychosis, Mania and Criminal Recidivism: Associations and Implications for Prevention. Harv Rev Psychiatry. 2020 May/Jun;28(3):179-202. doi: 10.1097/HRP.0000000000000251. PMID 32251070
- [Background] Elbogen EB, Johnson SC. The intricate link between violence and mental disorder: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Arch Gen Psychiatry. 2009 Feb;66(2):152-61. doi: 10.1001/archgenpsychiatry.2008.537. PMID 19188537
- [Background] Fazel S, Hayes AJ, Bartellas K, Clerici M, Trestman R. Mental health of prisoners: prevalence, adverse outcomes, and interventions. Lancet Psychiatry. 2016 Sep;3(9):871-81. doi: 10.1016/S2215-0366(16)30142-0. Epub 2016 Jul 14. PMID 27426440
- [Background] Ahonen L, Loeber R, Brent DA. The Association Between Serious Mental Health Problems and Violence: Some Common Assumptions and Misconceptions. Trauma Violence Abuse. 2019 Dec;20(5):613-625. doi: 10.1177/1524838017726423. Epub 2017 Aug 23. PMID 29333994
- [Background] Skjaervo I, Skurtveit S, Clausen T, Bukten A. Substance use pattern, self-control and social network are associated with crime in a substance-using population. Drug Alcohol Rev. 2017 Mar;36(2):245-252. doi: 10.1111/dar.12406. Epub 2016 May 4. PMID 27147068
- [Background] Mundt AP, Baranyi G. The Unhappy Mental Health Triad: Comorbid Severe Mental Illnesses, Personality Disorders, and Substance Use Disorders in Prison Populations. Front Psychiatry. 2020 Aug 14;11:804. doi: 10.3389/fpsyt.2020.00804. eCollection 2020. PMID 32922316
- [Background] Davison S, Janca A. Personality disorder and criminal behaviour: what is the nature of the relationship? Curr Opin Psychiatry. 2012 Jan;25(1):39-45. doi: 10.1097/YCO.0b013e32834d18f0. PMID 22156936
- [Background] Swanson JW, Holzer CE 3rd, Ganju VK, Jono RT. Violence and psychiatric disorder in the community: evidence from the Epidemiologic Catchment Area surveys. Hosp Community Psychiatry. 1990 Jul;41(7):761-70. doi: 10.1176/ps.41.7.761. PMID 2142118
- [Background] Fischer SN, Shinn M, Shrout P, Tsemberis S. Homelessness, mental illness, and criminal activity: examining patterns over time. Am J Community Psychol. 2008 Dec;42(3-4):251-65. doi: 10.1007/s10464-008-9210-z. PMID 18956238
- [Background] Coker KL, Smith PH, Westphal A, Zonana HV, McKee SA. Crime and psychiatric disorders among youth in the US population: an analysis of the National Comorbidity Survey-Adolescent Supplement. J Am Acad Child Adolesc Psychiatry. 2014 Aug;53(8):888-98, 898.e1-2. doi: 10.1016/j.jaac.2014.05.007. Epub 2014 Jun 12. PMID 25062596
- [Background] Moffitt TE. Adolescence-limited and life-course-persistent antisocial behavior: a developmental taxonomy. Psychol Rev. 1993 Oct;100(4):674-701. PMID 8255953
- [Background] Kalvin CB, Bierman KL. Child and adolescent risk factors that differentially predict violent versus nonviolent crime. Aggress Behav. 2017 Nov;43(6):568-577. doi: 10.1002/ab.21715. Epub 2017 Jun 8. PMID 28597509
- [Background] Costello EJ, Maughan B. Annual research review: Optimal outcomes of child and adolescent mental illness. J Child Psychol Psychiatry. 2015 Mar;56(3):324-41. doi: 10.1111/jcpp.12371. Epub 2014 Dec 12. PMID 25496295